CLINICAL TRIAL: NCT06038006
Title: A Clinical Trial Evaluating the Effectiveness and Safety of a Millimeter-Wave Radar Based Sleep Respiratory Monitoring System
Brief Title: A Clinical Trial Evaluating the Effectiveness and Safety of a mmWave Radar Based Sleep Respiratory Monitoring System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changsha Tsingray Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Beijing Tsingray Technology Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20221128
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Sleep Breathing Disorders

STUDY DESIGN:
Masking Description: During this study, results of the radar-based Sleep Respiratory Monitoring System are not known by the investigator and outcomes assessor, including the personnel who scores PSG.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): The only arm containing participants of this study.
  Interventions: Diagnostic Test: Sleep Respiratory Monitoring System

INTERVENTIONS:
Diagnostic Test: Sleep Respiratory Monitoring System — Millimeter-Wave radar-based Sleep Respiratory Monitoring System to be used on each participant undergoing PSG

SUMMARY:
This study compares the diagnostic capability of a millimeter-wave radar-based Sleep Respiratory Monitoring System to the gold standard polysomnography.

DETAILED DESCRIPTION:
The gold standard for the diagnosis of sleep breathing disorders is polysomnography (PSG), which requires contact sensors, in-lab monitoring and manual scoring by experts, limiting the comfortability of patients and accessibility of diagnosis. A novel contactless millimeter-wave radar-based Sleep Respiratory Monitoring System is developed, in order to assist sleep staging and the diagnosis of sleep breathing disorders.

The Sleep Respiratory Monitoring System is capable of collecting, recording, storing and analyzing breathing, heartbeat, spatial distribution of full-body movements, etc. via a millimeter-wave radar, and oxygen saturation, pulse, etc. via a pulse oximeter. A dedicated algorithm enables the system to detect respiratory events and estimate sleep stages based on the collected data. The device and algorithms are to be validated in this study by comparison with PSG.

ELIGIBILITY:
Inclusion Criteria:

* Participants is 18 years of age or older.
* Participants is willing to undergo overnight polysomnography and Sleep Respiratory Monitoring System testing.

Exclusion Criteria:

* Participants with severe cardiovascular and cerebrovascular diseases, severe liver, kidney, and lung dysfunction.
* Participants with unstable respiratory diseases, or other diseases in acute phase.
* Long-term or current use of barbiturates, benzodiazepines, sedatives and other drugs that may affect sleep.
* Participants that undergo CPAP treatment during the night of the trial.
* Participants with other sleep disorders, e.g. insomnia.
* Participants with mental disorders.
* Participants that refuse to sign informed consents.
* Participants unable to cooperate with medical examination.
* Participants excluded in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Sensitivity (AHI≥5) of Sleep Respiratory Monitoring System (SRMS) Compared with Polysomnography (PSG) | Day 1
  The proportion of participants with Apnea Hypopnea Index (AHI) ≥ 5 events per hour according to SRMS in participants with AHI ≥ 5 events per hour according to PSG scored with American Academy of Sleep Medicine (AASM) v2.6 Guidelines. The point estimation of diagnostic sensitivity of SRMS will be compared to the threshold of 0.8, with the half width of 95% confidence interval being no more than 0.1.
Diagnostic Sensitivity (AHI≥15) of Sleep Respiratory Monitoring System (SRMS) Compared with Polysomnography (PSG) | Day 1
  The proportion of participants with Apnea Hypopnea Index (AHI) ≥ 15 events per hour according to SRMS in participants with AHI ≥ 15 events per hour according to PSG scored with American Academy of Sleep Medicine (AASM) v2.6 Guidelines. The point estimation of diagnostic sensitivity of SRMS will be compared to the threshold of 0.8, with the half width of 95% confidence interval being no more than 0.1.
Diagnostic Sensitivity (AHI≥30) of Sleep Respiratory Monitoring System (SRMS) Compared with Polysomnography (PSG) | Day 1
  The proportion of participants with Apnea Hypopnea Index (AHI) ≥ 30 events per hour according to SRMS in participants with AHI ≥ 30 events per hour according to PSG scored with American Academy of Sleep Medicine (AASM) v2.6 Guidelines. The point estimation of diagnostic sensitivity of SRMS will be compared to the threshold of 0.8, with the half width of 95% confidence interval being no more than 0.1.
Diagnostic Specificity (AHI≥5) of Sleep Respiratory Monitoring System (SRMS) Compared with Polysomnography (PSG) | Day 1
  The proportion of participants with Apnea Hypopnea Index (AHI) < 5 events per hour according to SRMS in participants with AHI < 5 events per hour according to PSG scored with American Academy of Sleep Medicine (AASM) v2.6 Guidelines. The point estimation of diagnostic specificity of SRMS will be compared to the threshold of 0.8, with the half width of 95% confidence interval being no more than 0.1.
Diagnostic Specificity (AHI≥15) of Sleep Respiratory Monitoring System (SRMS) Compared with Polysomnography (PSG) | Day 1
  The proportion of participants with Apnea Hypopnea Index (AHI) < 15 events per hour according to SRMS in participants with AHI < 15 events per hour according to PSG scored with American Academy of Sleep Medicine (AASM) v2.6 Guidelines. The point estimation of diagnostic specificity of SRMS will be compared to the threshold of 0.8, with the half width of 95% confidence interval being no more than 0.1.
Diagnostic Specificity (AHI≥30) of Sleep Respiratory Monitoring System (SRMS) Compared with Polysomnography (PSG) | Day 1
  The proportion of participants with Apnea Hypopnea Index (AHI) < 30 events per hour according to SRMS in participants with AHI < 30 events per hour according to PSG scored with American Academy of Sleep Medicine (AASM) v2.6 Guidelines. The point estimation of diagnostic specificity of SRMS will be compared to the threshold of 0.8, with the half width of 95% confidence interval being no more than 0.1.

SECONDARY OUTCOMES:
Intra-Class Correlation Coefficient (ICC) of Apnea Hypopnea Index (AHI) | Day 1
  ICC between AHI according to Sleep Respiratory Monitoring System (SRMS) and AHI according to Polysomnography (PSG), using one-way random effects model.
Intra-Class Correlation Coefficient (ICC) of Total Sleep Time (TST) | Day 1
  ICC between TST according to Sleep Respiratory Monitoring System (SRMS) and TST according to Polysomnography (PSG), using one-way random effects model.
Intra-Class Correlation Coefficient (ICC) of Deep Sleep Proportion | Day 1
  ICC between the proportion of deep sleep time in total sleep time (TST) according to Sleep Respiratory Monitoring System (SRMS) and the proportion of stage N3 sleep time in TST according to Polysomnography (PSG), using one-way random effects model.
Intra-Class Correlation Coefficient (ICC) of Light Sleep Proportion | Day 1
  ICC between the proportion of light sleep time in total sleep time (TST) according to Sleep Respiratory Monitoring System (SRMS) and the proportion of stage N1 sleep time plus stage N2 sleep time in TST according to Polysomnography (PSG), using one-way random effects model.
Intra-Class Correlation Coefficient (ICC) of Rapid Eye Movement (REM) Sleep Proportion | Day 1
  ICC between the proportion of REM sleep time in total sleep time (TST) according to Sleep Respiratory Monitoring System (SRMS) and the proportion of stage R sleep time in TST according to Polysomnography (PSG), using one-way random effects model.

CONTACTS AND LOCATIONS:
Overall Officials: Shankai Yin, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li CY, Wang W, Huang WJ, Xu HH, Yi HL, Guan J, Li G, Yin SK. [Diagnosis of obstructive sleep apnea by a new radar device: a parallel controlled study evaluating agreement with polysomnographic monitoring]. Zhonghua Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2024 Aug 7;59(8):857-863. doi: 10.3760/cma.j.cn115330-20231204-00267. Chinese. PMID 39193596